CLINICAL TRIAL: NCT01142128
Title: A Randomized, Single Site, Double Blind, Fixed Dose, Cross Over Study of Viokase 16, Viokase16 Plus Nexium and Nexium Alone in the Reduction of Abdominal Pain in Patients With Chronic Pancreatitis
Brief Title: Viokase 16, Viokase16 Plus Nexium and Nexium Alone
Acronym: AZ
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Viokase was taken off market during study and remained off over a year.
Sponsor: University of Florida (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: D.9612.L00058
Record Dates: First submitted 2010-06-09; First posted 2010-06-11 (Estimated); Results first posted 2013-02-21 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Chronic Pancreatitis
MeSH Terms: conditions — Pancreatitis, Chronic | interventions — Esomeprazole; Pancrelipase

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Nexium alone (Active Comparator): Nexium alone is given for one month to be compared to a placebo to Nexium, Viokase 16 plus Nexium and Viokase 16 plus a placebo to Nexium
  Interventions: Drug: Nexium (esomeprazole magnesium)
- Placebo to Nexium, alone (Placebo Comparator): Placebo to Nexium is given instead of Nexium for one month. This will be compared to the Nexium alone, Viokase 16 plus Nexium and Viokase 16 plus placebo to Nexium
  Interventions: Drug: Placebo to Nexium
- Viokase 16 (pancrelipase) + Nexium (Active Comparator): Viokase 16 (pancrelipase) + Nexium capsules are given per day for one month with the addition of esomeprazole magnesium, one 40mg capsule per day for one month.
  Interventions: Drug: Viokase 16 (pancrelipase) + Nexium
- Viokase 16 + placebo to Nexium (Placebo Comparator): Viokase 16 is given with a placebo to Nexium for one month to be compared against Viokase 16 plus Nexium, Nexium alone and Placebo to Nexium alone
  Interventions: Drug: Viokase 16 + placebo to Nexium

INTERVENTIONS:
Drug: Nexium (esomeprazole magnesium) — one 40 mg capsule per day for one month
  Other Names: Nexium
  Arms: Nexium alone
Drug: Placebo to Nexium — one capsule per day for one month
  Arms: Placebo to Nexium, alone
Drug: Viokase 16 (pancrelipase) + Nexium — Viokase 16 (pancrelipase) + Nexium capsules are given per day for one month with the addition of esomeprazole magnesium, one 40mg capsule per day for one month
  Arms: Viokase 16 (pancrelipase) + Nexium
Drug: Viokase 16 + placebo to Nexium — Viokase 16 pancrelipase tablets are given per day for one month with one capsule of placebo to esomeprazole magnesium, one per day for one month
  Arms: Viokase 16 + placebo to Nexium

SUMMARY:
Our primary hypothesis is that the addition of Nexium to Viokase 16 will decrease the chronic abdominal pain in patients with small duct chronic pancreatitis in a superior fashion compared to Viokase 16 plus placebo or to Nexium alone. A secondary hypothesis would be an increase in quality of life. Our objective is to elucidate the role of Nexium in the control of pancreatic pain, quality of life, and narcotic usage alone or when added to Viokase 16. Our endpoints are the reduction of abdominal pain, decreased pain medication usage, decreased ER visits and decreased hospital admissions for abdominal pain.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females age 18 to 75 years inclusive. Female subjects of child bearing potential or less than two years post-menopausal must use a medically acceptable form of birth control or barrier method and have a negative pregnancy test prior to entry into study.
2. History of abdominal pain associated with chronic pancreatitis
3. Evidence of chronic pancreatitis as manifested by an abnormal secretin test, calcification of the pancreas on plain film, an abnormal CT showing a dilated pancreatic duct and/or atrophy, an abnormal Endoscopicretrogradecholangeopancreatography (ERCP), or diffuse changes on Endoscopic Ultrasound (EUS), fecal elastase > 100ug/g stool, or serum trypsinogen > 20ng/ml

   -

Exclusion Criteria:

1. Subjects on enzyme therapy within the last 14 days, proton pump inhibitor (PPI)within the last 7 days, or octreotide within 48 hours.
2. Subjects with known hypersensitivity to pork or exogenous or pancreatic enzymes.
3. Female subjects who are pregnant or lactating
4. Subject use of enzyme therapy other than that called for in this study
5. Subject use of therapeutic amounts of antacids or H2 receptor antagonists during the course of the study.
6. Past history of documented steatorrhea by 72 hour fecal fat determination or current history consistent with steatorrhea -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-02; Primary Completion 2011-12 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip P Toskes, M.D., Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The dates of the recruitment period were February 2009 through January 2010. Subjects recruited at the University of Florida and the Shands Hospital. Recruited a total of 12 subjects. Enrollment was slow due to subjects not wanting to come off their medications, this was unanticipated.
Pre-assignment Details: A total of 12 participants were consented to the study, however, 4 participants were never randomized to the study. Prior to randomization, subjects were off all enzymes and proton pump inhibitor's (PPI's) for 14 days.
Groups:
- All Participants: Participants received one of four interventions in a randomized crossover design:
  1. Nexium Alone: Nexium alone is given for one month to be compared to a placebo to Nexium, Viokase 16 plus Nexium and Viokase 16 plus a placebo to Nexium
  2. Placebo to Nexium, Alone: Placebo to Nexium is given instead of Nexium for one month. This will be compared to the Nexium alone, Viokase 16 plus Nexium and Viokase 16 plus placebo to Nexium
  3. Viokase 16 Plus Nexium: Viokase 16 is given with Nexium for one month to be compared against Nexium alone, Placebo to Nexium alone and Viokase 16 plus placebo to Nexium
  4. Viokase 16 Plus Placebo to Nexium: Viokase 16 is given with a placebo to Nexium for one month to be compared against Viokase 16 plus Nexium, Nexium alone and Placebo to Nexium alone
Period: Overall Study
Arm/Group | All Participants
Started | 8
Nexium Alone | 3
Placebo to Nexium, Alone | 3
Viokase 16 Plus Nexium | 2
Viokase 16 Plus Placebo to Nexium | 0
Completed | 4
Not Completed | 4
Not completed — Physician Decision | 1
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- Viokase 16 Plus Nexium: Viokase 16 is given with Nexium for one month to be compared against Nexium alone, Placebo to Nexium alone and Viokase 16 plus placebo to Nexium
- Viokase 16 Plus Placebo to Nexium: Viokase 16 is given with a placebo to Nexium for one month to be compared against Viokase 16 plus Nexium, Nexium alone and Placebo to Nexium alone
- Total: Total of all reporting groups
Arm/Group | Nexium Alone | Placebo to Nexium, Alone | Viokase 16 Plus Nexium | Viokase 16 Plus Placebo to Nexium | Total
Number analyzed (Participants) | 3 | 3 | 2 | 0 | 8
Age Categorical [Number; unit: participants]
  <=18 years | 0 | 0 | 0 |  | 0
  Between 18 and 65 years | 3 | 2 | 2 |  | 7
  >=65 years | 0 | 1 | 0 |  | 1
Gender [Number; unit: participants]
  Female | 1 | 2 | 1 |  | 4
  Male | 2 | 1 | 1 |  | 4
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 2 |  | 8

OUTCOME MEASURES:

1. Primary Outcome: Reduction of Abdominal Pain for Participants Taking Nexium Alone.
Description: To elucidate the role of Viokase 16 and Nexium in the control of pancreatic pain
Time Frame: 4 months
Population: Analysis was not able to be done due to the small sample size.
Groups:
- Nexium Alone: Viokase 16 is given with Nexium for one month to be compared against Nexium alone, Placebo to Nexium alone and Viokase 16 plus placebo to Nexium
Arm/Group | Nexium Alone
Number analyzed (Participants) | 0

2. Primary Outcome: Reduction of Abdominal Pain for Participants Taking Placebo to Nexium
Description: To elucidate the role of Viokase 16 and Nexium in the control of pancreatic pain
Time Frame: 4 months
Population: Analysis was not able to be done due to the small sample size.
Groups:
- Placebo to Nexium, Alone: Viokase 16 is given with Nexium for one month to be compared against Nexium alone, Placebo to Nexium alone and Viokase 16 plus placebo to Nexium
Arm/Group | Placebo to Nexium, Alone
Number analyzed (Participants) | 0

3. Primary Outcome: Reduction of Abdominal Pain in Participants Taking Viokase 16 Plus Nexium
Description: To elucidate the role of Viokase 16 and Nexium in the control of pancreatic pain
Time Frame: 4 months
Population: Analysis was not able to be done due to the small sample size.
Arm/Group | Viokase 16 Plus Nexium
Number analyzed (Participants) | 0

4. Primary Outcome: Reduction of Abdominal Pain in Participants Taking Viokase 16 Plus Placebo.
Description: To elucidate the role of Viokase 16 and Nexium in the control of pancreatic pain
Time Frame: 4 months
Population: Analysis was not able to be done due to the small sample size.
Groups:
- Viokase 16 Plus Placebo to Nexium: Viokase 16 is given with Nexium for one month to be compared against Nexium alone, Placebo to Nexium alone and Viokase 16 plus placebo to Nexium
Arm/Group | Viokase 16 Plus Placebo to Nexium
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from 03/02/2009 until 08/15/2010
Arm/Group | Nexium Alone | Placebo to Nexium, Alone | Viokase 16 Plus Nexium | Viokase 16 Plus Placebo to Nexium
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 0/2 | 0/0
Other Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 0/2 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nexium Alone (N=3) | Placebo to Nexium, Alone (N=3) | Viokase 16 Plus Nexium (N=2) | Viokase 16 Plus Placebo to Nexium (N=0)
GI Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nexium Alone (N=3) | Placebo to Nexium, Alone (N=3) | Viokase 16 Plus Nexium (N=2) | Viokase 16 Plus Placebo to Nexium (N=0)
Elevated Liver Enzymes (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No